CLINICAL TRIAL: NCT03986606
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of PSB205 in Patients With Relapsed/Refractory Solid Tumors
Brief Title: A Study of PSB205 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Puget Sound Biotherapeutics (dba Sound Biologics) (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSB205-001
Record Dates: First submitted 2019-06-04; First posted 2019-06-14 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Neoplasm Malignant
Keywords: neoplasm; checkpoint inhibitor; combination; immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Dose Escalation and Expansion Study of PSB205 (Experimental): Part 1 (Dose escalation): PSB205 will be administered in sequential cohorts of 3 to 6 subjects each receiving 1 of 5 doses of PSB205 on day 1 of every 21-day cycle (3 weeks) via IV infusion using a standard 3+3 dose escalation design. Dose escalation will continue until an MTD is reached.
  Part 2 (Dose Expansion): The clinical anti-tumor effects of PSB205 will be tested at the recommended Phase 2 dose (RP2D) determined during the dose-escalation phase in subjects from three different solid tumor cohorts.
  Interventions: Biological: PSB205

INTERVENTIONS:
Biological: PSB205 — PSB205 is a bi-functional product that has been engineered to contain two unique monoclonal antibodies.

SUMMARY:
This is an open-label, multicenter, Phase 1, ascending dose escalation study of PSB205 in subjects with advanced solid tumors. The study will be conducted in 2 parts. Part 1 of the study will be a dose escalation evaluation to determine the maximum tolerated dose (MTD) and to establish a recommended Phase 2 dose (RP2D) of PSB205. This study purpose is to describe the safety and tolerability, to assess Pharmacokinetics (PK) and immunogenicity, and to preliminarily assess the anti-tumor activity of PSB205 in subjects with solid tumors. Part 2 of the study will further evaluate the RP2D in 3 distinct tumor cohorts of approximately 12 subjects each.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2. Inclusion of subjects with an ECOG performance status of 2 should be discussed and is at the discretion of the sponsor's medical monitor and the investigator.
* Life expectancy of ≥3 months.
* Female subjects who are not pregnant or breastfeeding, 1 year postmenopausal, or surgically sterile and males even if surgically sterilized that Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.
* Suitable venous access for the study-required blood sampling, including PK and Pharmacodynamic sampling.

  1. To be enrolled in Part 1 (Dose escalation), subjects must have:

     1. Histologically confirmed diagnosis of advanced solid tumor and preferably radiographically or clinically measurable disease. Subjects with non-measurable, evaluable disease are permitted
     2. One or more prior lines of therapy . No curative options and progressed on or following standard of care therapy (SOC).
  2. To be enrolled in Part 2 (Dose expansion), subjects must have:

     1. Histologically confirmed diagnosis of advanced solid tumor of the following types, and radiographically or clinically measurable disease, one or more prior lines of therapy, no curative options and progressed on or following SOC.
     2. Squamous cell carcinomas- squamous non-small cell lung cancer (NSCLC) or squamous cell carcinoma of the head and neck (HNSCC)
     3. Locally advanced or metastatic gastric or gastroesophageal carcinoma
     4. Advanced or metastatic renal cell Carcinoma (clear cell, papillary, other)
     5. MSI-high colon carcinoma
     6. Small cell lung cancer
     7. Advanced urothelial cancer
     8. Metastatic melanoma I. Advanced soft-tissue or bone sarcoma

Exclusion Criteria:

1. Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
2. Grade 3 or Grade 4 irAEs related to prior cancer immunotherapy.
3. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression. Subjects previously treated central nervous system metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 14 days prior to first dose of study drug are permitted to enroll.
4. Hypertension unable to be controlled to ≤Grade 2 with medication.
5. Any condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before first dose of study drug. Corticosteroids for topical use, nasal spray, and inhaled steroids are allowed. Systemic corticosteroids for prophylaxis of contrast allergy are permitted.
6. Prior treatment with a CTLA-4 inhibitor in combination with a PD-1 or PD-L1 inhibitor.
7. Systemic anti-cancer treatment (including investigational agents). This includes radiotherapy <2 weeks before the first dose of study drug, ≤4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T cell engaging agents; (≤8 weeks for cell-based therapy or anti-tumor vaccine) or have not recovered from acute toxic effects from prior chemotherapy and radiotherapy.
8. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
9. Systemic infection requiring IV antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
10. Subjects with a history of organ transplant.
11. Hepatitis B surface antigen-positive or known or suspected active hepatitis C infection.
12. Known human immunodeficiency virus (HIV) positive.
13. Subjects with any of the following cardiovascular conditions are excluded:

    1. Acute myocardial infarction within 6 months before first dose of study drug.
    2. Current or history of New York Heart Association Class III or IV heart failure.
    3. Evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
14. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
15. Subject has a history of alcoholism or drug abuse within the past 6 months.
16. Vaccinations within 4 weeks of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-07-28 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 28 days
  Safety and tolerability, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Next Oncology, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No